CLINICAL TRIAL: NCT01347619
Title: iADAPT: Off Label Use of Antipsychotics in the Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Qualidigm (Industry); Omnicare Clinical Research (Industry)
Responsible Party: Principal Investigator, Jerry Gurwitz, Executive Director, Meyers Primary Care Inst., University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13902
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Off-label Use of Atypical Antipsychotic Drugs
Keywords: Comparative Effectiveness Research Summary Guide (CERSG); anti-psychotic use; Nursing Home; Long-term care; Qualitative assessment of influences on CERSG adoption in NH; Development of toolkit of CERSG-based products for NHs; Evaluation of 3 implementation strategies of the toolkit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1. Toolkit only with Web Access (Active Comparator): NHs in this arm will receive the toolkit only and web access to the materials.
  Interventions: Other: Toolkit only with Web Access to Online Version
- Arm 2.Toolkit, Audit/Feedback, Education (Active Comparator): NHs in the second arm will receive the toolkit, web access, periodic audit and feedback reports of antipsychotic prescribing to NH leadership, and faxed educational messages adapted from the AHRQ atypical antipsychotic CERSG to prescribers.
  Interventions: Other: Toolkit, Periodic Audit/Feedback, Educational Messages
- Arm 3. All above plus academic detailing (Active Comparator): NHs in the third arm will receive the previous items plus face-to-face academic detailing.
  Interventions: Other: Items in Arm 2 plus Academic Detailing Program

INTERVENTIONS:
Other: Toolkit only with Web Access to Online Version — NHs in this arm will receive a letter announcing the availability of an atypical antipsychotic toolkit within the facility and online at the Qualidigm website. The letter will be sent to the NH administrator, Director of Nursing, and Medical Director of each facility by Qualidigm. It will state that the toolkit is designed to provide NH staff, including prescribers, leadership, nursing staff, and patients' families with information about the use, risks and costs of atypical antipsychotics in the NH setting.
  Arms: Arm 1. Toolkit only with Web Access
Other: Toolkit, Periodic Audit/Feedback, Educational Messages — Providing healthcare professionals with data about their performance (audit and feedback) may help improve their practice. It is more effective when clinicians previously agree to review their practice. We will use an adaptation of a "Medicaid Utilization Report" developed by AM Hamer. This report will show current atypical antipsychotic prescribing rates in the NH, with comparisons to state and national levels, and information regarding summary evidence for atypical antipsychotics from the AHRQ atypical antipsychotic CERSG. Reports will be sent to the NH administrator, Director of Nursing, and Medical Director of the facilities randomized to the moderate intensity arm on an every 4-month basis.
  Arms: Arm 2.Toolkit, Audit/Feedback, Education
Other: Items in Arm 2 plus Academic Detailing Program — This arm will receive the same information, toolkit, letters, and audit and feedback reports distributed to homes in the moderate-intensity arm. In addition, two visits to the NH will be scheduled by a pharmacist educator specially trained in the pharmacology of atypical antipsychotics, and communication techniques. Staff will be provided with up-to-date, unbiased information about antipsychotic use in NHs based on the AHRQ CER Review product adaptations. The educator will deliver targeted messages relevant to each stakeholder regarding roles in decision-making around the use atypical antipsychotic therapy in the NH setting. Each NH will receive up to two visits over the course of the 12-month intervention period.
  Arms: Arm 3. All above plus academic detailing

SUMMARY:
The investigators propose to evaluate the effectiveness of 3 different methods to promote the dissemination and adoption of evidenced-based review guides into the nursing home setting. Specifically, the investigators will adapt Comparative Effectiveness Research (CER) Review products developed by the Agency for Healthcare Research and Quality (AHRQ), specifically related to off-label use of atypical antipsychotic drugs, to improve their penetration into practice in the nursing home (NH) setting.

The investigators propose the following specific aims:

AIM 1: NEEDS ASSESSMENT To conduct a needs assessment for the NH setting relevant to the AHRQ Comparative Effectiveness Research Summary Guide (CERSG) entitled "Off-Label Use of Atypical Antipsychotic Drugs." The assessment will identify: (a) interest in and barriers to the use of the AHRQ atypical antipsychotic CERSG in the NH setting; (b) the key audiences and stakeholders that influence atypical antipsychotic drug use in NHs; and (c) approaches to integrating comparative effectiveness research products into the NH setting.

AIM 2: PRODUCTION OF THE TOOLKIT Guided by the needs assessment, the investigators will produce a toolkit containing tailored CERSG-based products targeting key audiences and stakeholders in the NH setting. The target audience(s) of the final CERSG-based products will be identified in Aim 1, and will potentially include: (a) facility leadership [NH administrator, Medical Director, Director of Nursing]; (b) prescribers and consultant pharmacists; (c) nursing staff [registered nurses, licensed practical nurses, and certified nurse assistants].

AIM 3: EVALUATING THE EFFECTIVENESS OF THE TOOLKIT To evaluate the effectiveness of the toolkit and three dissemination strategies using a matched, cluster randomized trial. NHs in the first arm will receive the toolkit only and web access to the materials; NHs in the second arm will receive the toolkit, web access, periodic audit and feedback reports of antipsychotic prescribing to NH leadership, and faxed educational messages adapted from the AHRQ atypical antipsychotic CERSG to prescribers; and NHs in the third arm will receive the previous items plus face-to-face academic detailing. Primary outcomes of the evaluation are the RE-AIM evaluation domains (reach, efficacy, adoption, implementation, and maintenance).The investigators will also include an assessment of facility-level changes in the use of atypical antipsychotic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Qualidigm-affiliated Nursing Home facilities in Connecticut who agree to participate.

Participants in this study will include residents and employees of participating nursing homes or residents within these nursing homes. All members of this study population will be 18 years or older.

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Aim 1 NEEDS ASSESSMENT - to describe interest in and barriers to the use of the AHRQ atypical antipsychotic CERSG | months 4-8
  Aim 1 - To conduct a needs assessment for the NH setting relevant to the AHRQ Comparative Effectiveness Research Summary Guide (CERSG) entitled "Off-Label Use of Atypical Antipsychotic Drugs." The assessment will identify: (a) interest in and barriers to the use of the AHRQ atypical antipsychotic CERSG; (b) the key audiences and stakeholders that influence atypical antipsychotic drug use in NHs; and (c) approaches to integrating comparative effectiveness research products into the NH setting
Aim 1 NEEDS ASSESSMENT - to describe the key audiences and stakeholders that influence atypical antipsychotic drug use in NHs | months 4-8
  Aim 1 - To conduct a needs assessment for the NH setting relevant to the AHRQ Comparative Effectiveness Research Summary Guide (CERSG) entitled "Off-Label Use of Atypical Antipsychotic Drugs." The assessment will identify: (a) interest in and barriers to the use of the AHRQ atypical antipsychotic CERSG; (b) the key audiences and stakeholders that influence atypical antipsychotic drug use in NHs; and (c) approaches to integrating comparative effectiveness research products into the NH setting.
Aim 1 NEEDS ASSESSMENT - to describe approaches to integrating comparative effectiveness research products into the NH setting | months 4-8
  Aim 1 - To conduct a needs assessment for the NH setting relevant to the AHRQ Comparative Effectiveness Research Summary Guide (CERSG) entitled "Off-Label Use of Atypical Antipsychotic Drugs." The assessment will identify: (a) interest in and barriers to the use of the AHRQ atypical antipsychotic CERSG; (b) the key audiences and stakeholders that influence atypical antipsychotic drug use in NHs; and (c) approaches to integrating comparative effectiveness research products into the NH setting.
Aim 2 - Guided by the needs assessment, we will produce a toolkit containing tailored CERSG-based products targeting key audiences and stakeholders in the NH setting. | months 9-12
  Aim 2 - Guided by the needs assessment, we will produce a toolkit containing tailored CERSG-based products targeting key audiences and stakeholders in the NH setting. The targets of the final CERSG-based products will be identified in Aim 1, and will potentially include: (a) facility leadership [NH administrator, Medical Director, Director of Nursing]; (b) prescribers and consultant pharmacists; (c) nursing staff [registered nurses, licensed practical nurses, and certified nurse assistants], and (d) residents and families.
Aim 3 - To evaluate the effectiveness of the toolkit and three dissemination strategies using a matched, cluster randomized trial | months 31-36
  Aim 3 - To evaluate the effectiveness of the toolkit and three dissemination strategies using a matched, cluster randomized trial. Primary outcomes of the evaluation are the RE-AIM evaluation domains (reach, efficacy, adoption, implementation, and maintenance).

CONTACTS AND LOCATIONS:
Overall Officials: Jerry H Gurwitz, MD, Principal Investigator — UMass Medical School
Locations (1):
- Qualidigm, Rocky Hill, Connecticut, United States

REFERENCES:
- [Result] Tjia J, Gurwitz JH, Briesacher BA. Challenge of changing nursing home prescribing culture. Am J Geriatr Pharmacother. 2012 Feb;10(1):37-46. doi: 10.1016/j.amjopharm.2011.12.005. Epub 2012 Jan 20. PMID 22264855
- [Result] Lemay CA, Mazor KM, Field TS, Donovan J, Kanaan A, Briesacher BA, Foy S, Harrold LR, Gurwitz JH, Tjia J. Knowledge of and perceived need for evidence-based education about antipsychotic medications among nursing home leadership and staff. J Am Med Dir Assoc. 2013 Dec;14(12):895-900. doi: 10.1016/j.jamda.2013.08.009. Epub 2013 Sep 24. PMID 24074962
- [Result] Briesacher BA, Tjia J, Field T, Peterson D, Gurwitz JH. Antipsychotic use among nursing home residents. JAMA. 2013 Feb 6;309(5):440-2. doi: 10.1001/jama.2012.211266. No abstract available. PMID 23385262
- [Result] Tjia J, Field T, Lemay C, Mazor K, Pandolfi M, Spenard A, Ho SY, Kanaan A, Donovan J, Gurwitz JH, Briesacher B. Antipsychotic use in nursing homes varies by psychiatric consultant. Med Care. 2014 Mar;52(3):267-71. doi: 10.1097/MLR.0000000000000076. PMID 24374410